CLINICAL TRIAL: NCT07081802
Title: the Effect of Perioperative Transcutaneous Electrical Acupoint Stimulation Combined With Traditional Chinese Medicine on Gastrointestinal Function Recovery in Abdominal Surgery Patients
Brief Title: Effect of Acupuncture and Herbal Medicine on Bowel Recovery After Abdominal Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Guang'anmen Hospital of China Academy of Chinese Medical Sciences (Other)
Collaborators: Second Affiliated Hospital of Nanchang University (Other); The First Hospital of Qinhuangdao (Other Government); Affiliated Hospital of Hebei University (Other); Handan Central Hospital (Other); Liaoning Cancer Hospital & Institute (Other)
Responsible Party: Principal Investigator, Quanda Liu, Chief Physician, Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025-037-KY-01
Record Dates: First submitted 2025-07-07; First posted 2025-07-23 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: ERAS; Traditional Chinese Medication (TCM)
MeSH Terms: interventions — dai-kenchu-to; ginger extract; Asian ginseng; Maltose

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TEAS + TCM + Prehabilitation + ERAS (Experimental): Experimental Group:
  TEAS:
  Administered once daily from the day of surgery until postoperative day 4. Each session lasts 30 minutes, except on the day of surgery, when treatment begins 30 minutes preoperatively and continues for 1 hour.
  Acupoints: ST36 (Zusanli), ST37 (Shangjuxu), PC6 (Neiguan), and LI4 (Hegu) Note: Intraoperatively, only bilateral ST36 and ST37 are stimulated due to anesthesia constraints.
  Parameters: Continuous wave at 10 Hz; intensity adjusted to elicit deqi sensation (heaviness, numbness, or soreness) within patient tolerance.
  Traditional Chinese Medicine (TCM):
  Intraoperative & Postoperative (up to day 4): Fixed prescription of Da Jian Zhong Tang Zanthoxyli Pericarpium (Sichuan Pepper) 3g, Zingiberis Rhizoma (Dried Ginger) 12g, Ginseng Radix et Rhizoma (Ginseng) 6g, Maltosum (Malt Sugar) 30g.
  All participants receive identical perioperative management and postoperative care, including prehabilitation and Enhanced Recovery After Surgery (ERAS) protocols.
  Interventions: Drug: Da Jian Zhong Tang (Zanthoxylum, Ginger, Ginseng, Maltose); Procedure: Transcutaneous Electrical Acupoint Stimulation (TEAS); Other: ERAS; Other: Multimodal Prehabilitation Program
- Prehabilitation + ERAS (Active Comparator): All participants receive identical perioperative management and postoperative care, including prehabilitation and Enhanced Recovery After Surgery (ERAS) protocols.
  Interventions: Other: ERAS; Other: Multimodal Prehabilitation Program

INTERVENTIONS:
Drug: Da Jian Zhong Tang (Zanthoxylum, Ginger, Ginseng, Maltose) — "Da Jian Zhong Tang (Zanthoxylum, Ginger, Ginseng, Maltose)was administered orally twice daily from preoperative day 3 to postoperative day 3. The decoction aims to warm the middle jiao and promote gastrointestinal recovery, with dose adjustments based on syndrome differentiation.
  Arms: TEAS + TCM + Prehabilitation + ERAS
Procedure: Transcutaneous Electrical Acupoint Stimulation (TEAS) — TEAS was delivered at acupoints ST36/ST37 (10Hz continuous wave, 30min/session) once daily from intraoperative day to postoperative day 4. On surgery day, stimulation started 30min preoperatively for 1 hour. Intensity was adjusted to elicit deqi sensation.
  Arms: TEAS + TCM + Prehabilitation + ERAS
Other: ERAS — "Standardized ERAS protocol included: (1) Preoperative carbohydrate loading; (2) Intraoperative goal-directed fluid therapy; (3) Minimally invasive surgery; (4) Multimodal opioid-sparing analgesia; (5) Early oral feeding (semi-liquid diet at 6h post-op); (6) Early ambulation (first mobilization at 8h post-op). Implemented by a multidisciplinary team.
  Other Names: Fast-Track Surgery
Other: Multimodal Prehabilitation Program — (1) Exercise: Daily aerobic/resistance training (30min, 5×/week); (2) Nutrition: High-protein diet (1.5g/kg/day) + oral supplements if needed; (3) Psychological Support: Cognitive-behavioral therapy sessions (2×/week). Tailored to individual patient risk profiles.

SUMMARY:
Protocol Summary Project Name:Effect of Perioperative TEAS Combined with TCM on Gastrointestinal Function Recovery in Abdominal Surgery Patients Research Objective:To evaluate the impact of perioperative TEAS combined with TCM on postoperative gastrointestinal function, pain, adverse reactions, hospital stay, and complications, as well as its safety, aiming to enrich the ERAS and prehabilitation theory and promote the integration of TCM in surgical practice.

Research Design:Prospective, randomized, open-label trial involving 148 abdominal surgery patients (Grade IV surgeries) randomly assigned 1:1 to the experimental group (TCM + TEAS + prehabilitation + ERAS) or the control group (prehabilitation + ERAS).

Total Cases:148 Case Selection

Inclusion Criteria:

1. Age 18-80, no severe gastrointestinal dysfunction;
2. Elective abdominal Grade IV surgeries (pancreas or colorectall surgeries) via open or laparoscopic methods;
3. Preoperative ASA classification I-III;
4. Signed informed consent.

Exclusion Criteria:

Severe comorbidities, skin abnormalities at acupoints, long-term use of gastrointestinal motility drugs, or other factors affecting the trial.

Elimination Criteria:

Poor compliance, significant missing data, or severe adverse events unrelated to the intervention.

Treatment Plan TEAS combined with TCM from the day of surgery to postoperative day 4, alongside prehabilitation and ERAS.

Efficacy Evaluation

Primary Outcomes:

Time to first flatus and defecation.

Secondary Outcomes:

Postoperative hospital stay, time to tolerate semi-liquid/solid food, nausea/vomiting, pain, bloating, first ambulation, 30-day readmission rate, WBC/CRP levels, and gastrin levels.

Safety Evaluation: Any adverse events. Statistical Methods Continuous variables expressed as mean (SD) or median (IQR); independent t-test for normal distributions. Categorical variables summarized as frequencies/percentages, analyzed using χ² or Fisher's exact test. Group differences reported as 95% CI and two-sided P-values (P < 0.05 significant). Preset subgroup analyses by surgery type and frailty.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged >18 years with no severe preoperative gastrointestinal dysfunction (e.g., no chronic gastrointestinal diseases such as long-term constipation or diarrhea).
* Scheduled abdominal Grade IV surgeries (limited to liver, gallbladder, pancreas, stomach, or intestinal procedures) performed via open or laparoscopic approach.
* Preoperative American Society of Anesthesiologists (ASA) Physical Status Classification of I-III.
* Patients and their families fully understand the study's purpose, methods, potential risks/benefits, and provide signed informed consent.

Exclusion Criteria:

* Comorbid severe systemic diseases.
* Local skin abnormalities at acupoints (e.g.,broken skin, infection, allergies, or scarring).
* Preoperative long-term use (>1 month) of gastrointestinal motility-affecting drugs (e.g., mosapride, domperidone) that cannot be discontinued, or allergies to TCM components/electrode materials.
* Psychiatric disorders or cognitive impairment rendering patients unable to comply with the study.

Elimination Criteria:

* Non-compliance with treatment protocols (e.g., receiving <80% of planned sessions).
* Significant missing data.
* Occurrence of severe adverse events unrelated to the study intervention.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-09-28 (Estimated)

PRIMARY OUTCOMES:
Time to First Defecation | Time to first defecation was recorded from the moment sugery finished until the first defecation occurred, with a maximum observation period of 4 days
  Defined as the interval from the end of surgery to the first observed bowel movement.
Time to first flatus | Time to first flatus was recorded from the moment sugery finished until the first flatus occurred, with a maximum observation period of 4 days
  Defined as the interval from the end of surgery to the first passage of gas.
Serological Markers | Measured preoperatively (day 1 before surgery) and on postoperative day 3.
  White blood cell (WBC) count and C-reactive protein (CRP)

SECONDARY OUTCOMES:
Postoperative Hospital Stay | Time to first defecation was recorded from the moment sugery finished until the first defecation occurred, with a maximum observation period of 4 days
  Postoperative hospital stay was defined as the duration from end of surgery to hospital discharge, measured in days
Time to Tolerate Semi-Liquid and Solid Foods | postoperative
  Defined as the interval from the end of surgery to the first successful intake of semi-liquid (e.g., congee, egg custard) or solid food without nausea, vomiting, or other gastrointestinal adverse reactions.
  Tolerance criteria: No nausea or vomiting within 4 hours after eating.
Postoperative Nausea and Vomiting (PONV) | postoperative day 1 to day 7
  Assessed daily from postoperative day 1 to day 7 using a VAS (0-100 mm), where 0 = "no nausea" and 100 = "worst possible nausea."
  The frequency of nausea/vomiting episodes was recorded (intervals >5 minutes counted as separate events).
Postoperative Pain | from postoperative day 1 to day 7
  Evaluated daily (days 1-7) using VAS (0-100), where 0 = "no pain" and 100 = "worst imaginable pain."
  Recorded at 8:00 AM for the preceding 24-hour period.
Time to First Ambulation | Time to first Ambulation was recorded from the moment sugery finished until the first Ambulation occurred, with a maximum observation period of 4 days
  Defined as the interval from the end of surgery to the first out-of-bed activity.
30-Day Readmission Rate | postoperative day 30
  The proportion of patients readmitted within 30 days after discharge due to surgery-related complications.
Serum gastrin levels | Preoperative day 1 Postoperative day 3 Postoperative day 7
  Assessed via ELISA or chemiluminescence at three time points:

IPD SHARING:
Plan to Share IPD: No